CLINICAL TRIAL: NCT06692998
Title: Comparison of the Efficacy of High and Low Level Laser Therapy in the Treatment of De Quervain's Tenosynovitis: a Randomized Controlled Trial
Brief Title: High and Low Level Laser Therapy in De Quervain's Tenosynovitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SADEQ
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: DeQuervain Tendinopathy
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HILT Group (Experimental): Patients will receive pulsed laser therapy using the HIRO 3 device (ASA Laser, Arcugnano, Italy) five times a week for 3 weeks, one session per day for a total of 15 sessions. The HILT device offers pulsed emission (1064 nm), very high peak power (3 kW), high fluence (energy density 360-1780 mJ/cm2), short duration (120-150 μs), average power of 10.5 W, low frequency (10-40 Hz), duty cycle of approximately 0.1%, a 0.5 cm diameter probe and a spot size of 0.2 cm. A standard handpiece equipped with fixed spacers is used to maintain the same distance from the skin. The 3-stage treatment program is planned to be applied to the 1st CMC joint area in each session.
  Interventions: Other: Rehabilitation
- LLLT Group (Active Comparator): The MLS Multiwave Locked System laser device will be used for the treatment (low level laser). The laser probe (1 cm in diameter) will be applied directly and perpendicularly and lightly in contact with the skin. LLLT for de quatrein will be applied twice per session. Once the probe will be held in contact with the skin (at the radial styloid) and the second time in scanning mode (approximately 1 inch long along the tendon sheath). The area to be treated will be divided into 1 cm square areas and the optimum anti-inflammatory dosage (3 J/cm) continuous output mode will be used
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Patients will do hand-wrist joint range of motion, stretching and strengthening exercises for 20 minutes once a day, under the supervision of the same physiotherapist.

SUMMARY:
The aim in this study was to compare the effects of high and low power laser treatments in the treatment of de Quervein tenosynovitis clinically and ultrasonographically.

DETAILED DESCRIPTION:
De Quervain's tenosynovitis is tenosynovitis of the abductor pollicis longus (APL) and extensor pollicis brevis (EPB) tendons. Conservative management includes nonsteroidal anti-inflammatory drugs, wrist and thumb immobilization, ultrasound, and low-level laser therapy (LLLT). According to early literature, low-level laser therapy and ultrasound therapy appear to produce similar biological effects in reducing inflammation and promoting tissue healing.

In a study low-power laser therapy was found to be effective compared to placebo in de Quervain's tenosynovitis.

In a study of 35 female patients, low-power laser therapy (LLLT) combined with a thumb-supported splint was not superior to splint alone in patients with de Quervain's tenosynovitis.

In a more recent study low-power laser therapy was found to be similarly effective to ultrasound therapy.

The investigators found no studies in the literature on the effect of high-power laser therapy. The aim in this study was to compare the effects of high and low power laser treatments in the treatment of de Quervein tenosynovitis clinically and ultrasonographically.

ELIGIBILITY:
Inclusion Criteria:

* Between18-65 years of age
* Wrist pain for more than 3 weeks
* Finkelstein test positive
* Ability to understand commands

Exclusion Criteria:

* Physical therapy, injections, or surgery in the upper extremity in the last 3 months
* Fracture or trauma in the upper extremity in the last 6 months
* Radiating pain due to cervical discopathy
* Infection, loss of sensation, metal implant in the treatment area
* Inflammatory rheumatic diseases
* NSAID use
* Pregnancy or planning pregnancy during treatment
* Malignancy
* Pathology in the wrist on radiograph

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Pain Scale (VAS) | Before treatment (T0), After tratment (3. week) (T1)
  Visual Pain Scale (VAS), which is easy to understand, apply and interpret, and provides valid and reliable data in a short time, is the most commonly used method in clinics. With a 100 mm visual linear scale, the patient is told that there is no pain at point 0, and that the most severe pain they have ever felt at point 100, and the patient is asked to put a mark on the point corresponding to their pain.
Ritchie Articular Index | Before treatment (T0), After tratment (3. week) (T1)
  It is an index developed for the numerical measurement of joint tenderness in patients with rheumatoid arthritis. It is the quantitative evaluation number of the patient's response to the discomfort experienced by the joint when exposed to pressure during passive movement of the joint. It is a 4-point scale; if there is no tenderness (0), the patient complains of pain (1), the patient complains of pain and is accompanied by patient irritation (2), and the patient withdraws with pain and irritation (3). As a result, the total score obtained by summing the clinical evaluation index items made with joint tenderness is recorded.
Finkelstein test | Before treatment (T0), After tratment (3. week) (T1)
  The Finkelstein test is the occurrence of wrist pain at the level of the radial styloid during ulnar deviation of the wrist with the thumb flexed into the palm and covered with the remaining fingers.
Jamar Dynamometer | Before treatment (T0), After tratment (3. week) (T1)
  Measurements will be made by sitting with the shoulder adducted and neutrally rotated, adjacent to the body, elbow 90 degrees flexed, wrist 0-30 degrees dorsiflexed and 0-15 degrees ulnar deviation, thumb up. Measurements will be repeated three times with 5-second intervals on the affected hand and the average of the three measurements will be recorded in kilograms. Finger grip strength will be assessed with the 'Jamar digital pinchmeter'.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand Questionnaire (QUICK DASH) | Before treatment (T0), After tratment (3. week) (T1)
  It is used to measure physical function and symptoms in patients with upper extremity musculoskeletal disorders.The questionnaire consists of a disability/symptom scale (11 items) and two optional scales: work (four items) and sports/performing arts (four items). Each item on the disability/symptom scale asks about pain intensity, activity-related pain, tingling, weakness and stiffness, difficulty moving, physical activity due to upper extremity problems, and the impact of upper extremity problems on social activities, work and sleep. Responses are given on a one-to-five scale, with each question scored from 1 to 5. From the item scores, scale scores are calculated, ranging from 0 (no disability) to 100 (most severe disability).
Ultrasonographic evaluation | Before treatment (T0), After tratment (3. week) (T1)
  Ultrasonographic evaluation for both wrists will be performed by the same physiatrist who is unaware of the participant's clinical data and group distribution using the Esaote My Lab 70 Vision USG device with a 7.5 MHz linear probe. The combined thickness of the APL and EPB sheaths will be measured. In addition, the presence of fluid and Doppler activity around the tendon will be assessed. Patients are assessed in a sitting position with both forearms placed on the patient's lap/thigh in a mid-prone position. The scanned area will extend from a few centimeters proximal to the radial styloid to the insertion of the tendons of the first compartment (distal end of the proximal phalanx). Transverse scans will be obtained for measurement of the tendon sheath at the level of the radial styloid.

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA ADAR, Ass. Prof., Principal Investigator — Afyonkarahisar Health Sciences University

IPD SHARING:
Plan to Share IPD: No